CLINICAL TRIAL: NCT04818008
Title: Measuring the Effect of Using the Arabic Otago Exercise Program on Falls and Falls-related Factors in People With Multiple Sclerosis
Brief Title: The Use of Arabic Otago Exercise Program in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Alia A. Alghwiri, Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: "11-2021"
Record Dates: First submitted 2021-01-28; First posted 2021-03-26 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
Keywords: Otago Exercise Program; Falls
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Program (Experimental): Patients will receive the Otago Exercise Program for 8 weeks plus health awareness videos about topics related to MS.
  Interventions: Other: Otago Exercise Program
- Control group (No Intervention): Patients will receive health awareness videos only about topics related to MS.

INTERVENTIONS:
Other: Otago Exercise Program — A Home-based Exercise Program to improve strength and balance and prevent falls.
  Arms: Otago Exercise Program

SUMMARY:
People with multiple sclerosis (MS) need exercise training programs throughout their life in order to prevent secondary complications of the disease. Coronavirus disease of 2019 (COVID-19) forced people with chronic disorders to stay at home in order to prevent the transmission of the virus. Therefore, people with MS now are facing a new challenge in going outside their home to perform their rehabilitation sessions. One of the solutions to keep them exercising is a home-based exercise program and one of the home exercise programs that are well validated in older adults is the Otago exercise program (OEP). Investigators suggest that the balance would improve and fall incidences would reduce using the OEP in people with MS compared to health awareness videos only.

50 participants with confirmed diagnosis of MS will be recruited in both groups. Using a randomized controlled trial this study aims to examine the effectiveness of the OEP compared to a control group that gets health awareness videos only on falls and falls-related factors in people with MS.

DETAILED DESCRIPTION:
Ethical consideration:

This study got the ethics approval from the deanship of scientific research ethical committee at University of Jordan. A consent form that contains the study procedures will be prepared and signed from all patients.

Design:

This will be a single blinded randomized controlled trial study with 2 groups. The treatment group will receive the OEP for 8 weeks plus health awareness videos about topics related to MS. The control group will receive only the same health awareness videos. The health awareness videos will be video-recorded by a health-care provider then sent to all participants on weekly basis.

Participants:

People with a confirmed diagnosis of MS will be approached via their society and social media.

Procedures:

This trial will be registered on "clinicaltrials.gov" registry prior to the conduction of the study. Patients will be screened for eligibility and interested individuals will be informed about the study details and sign the informed consent.

All participants will be invited to University of Jordan for the baseline and end of program assessment. Demographics (age, gender, marital status, educational level) and health-related information (weight in kilograms and height in meters to be combined to report BMI in kg/m^2) and (caffeine consumption, smoking, present medical history, and Expanded Disability Status Scale score) will be gathered before going through the study measurements as baseline assessment by a licensed physical therapist (PT). The study measurements include fall history, chair balance test, four test balance scale, the Modified Fatigue Impact Scale (MFIS), Hand Held Dynamometer (HHD) for quadriceps muscle, Timed-Up and go (TUG), the Falls Efficacy Scale-International (FES-I), the Pittsburgh Sleep Quality Index (PSQI), the Hospital Anxiety and Depression Scale (HADS), the Medical Outcomes Study Short Form 12 (SF-12), and the Montreal Cognitive Assessment (MoCA).

Afterward, participants will be randomly allocated to the treatment or control groups using a computer-generated software. After 8 weeks, each participant in both groups will be reassessed using the same measurements used at the baseline assessment. Follow up questions about falls will be asked in 6 and 12 months post-treatment.

Participants in the treatment group will be visited at their homes each 2 weeks. In the first visit, the following steps will be conducted: (1) establish a good working relationship with the participant, (2) explain the rationale for the program, (3) prescribe a set of exercises from the OEP booklet and encourage the person to become familiar with the instructions for each exercise, and (4) if possible, introduce a safe walking plan. Participants in the treatment group will progress their exercises each 2 weeks to complete the 4 levels of OEP during the 8 weeks according to the instructions of the OEP. The PT will call participants weekly to make sure they are doing their exercises and to record any adverse events like relapse or falling.

Participants in the control group will be provided with health awareness videos about topics related to MS and inform them to avoid engagement in any exercise programs during the period of the study. Participants will be called weekly to make sure they adhere to the instructions.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years and older.
2. Both genders
3. All types of multiple sclerosis.
4. Independent in ambulation even with the use of an assistive device.
5. An Expanded Disability Status Scale (EDSS) score ≤ 6.5.

Exclusion Criteria:

1. The diagnosis of other neurological or musculoskeletal disorders that affect balance.
2. If the patient had a relapse within that last four weeks.
3. wheelchair users.
4. If the patient is engaged in any exercise program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of falls | 2 months post intervention.
  The effect of the intervention on the incidence of falls.
Incidence of falls | 6 months post intervention.
  The effect of the intervention on the incidence of falls.
Incidence of falls | 12 months post intervention.
  The effect of the intervention on the incidence of falls.

SECONDARY OUTCOMES:
Fear of Falling (using the Falls Efficacy Scale-International ) | 2 months post intervention.
  The effect of the intervention on fear of falling. The total score ranges between 16 and 64 with a higher score indicates greater fear of falling (worse).
Balance (using Chair balance test and Four test balance scale) | 2 months post intervention.
  The effect of the intervention on balance. The time taken to conduct these balance tasks are timed using a stopwatch. The longer the time taken by the patient to perform the tasks, the worse the balance. There is no minimum or maximum scores for these tests.
Mobility (using Timed-Up and go) | 2 months post intervention.
  The effect of the intervention on mobility. This assessments of mobility is timed out using a stopwatch.
Quadriceps strength (using a dynamometer) | 2 months post intervention.
  The effect of the intervention on quadriceps strength. The strength of quadriceps will be assessed using a dynamometer in kilograms.
The severity of fatigue (using Modified Fatigue Impact Scale) | 2 months post intervention.
  The effect of the intervention on the severity of fatigue. The total score ranges from 0 to 84 with a higher score indicates greater severity of fatigue symptoms (worse).
the Quality of sleep (Using Pittsburgh Sleep Quality Index) | 2 months post intervention.
  The effect of the intervention on the Quality of sleep. The total score ranges from 0 to 21 with a higher score indicates poor quality of sleep (worse).
the severity of Anxiety and Depression (using Hospital Anxiety and Depression Scale) | 2 months post intervention.
  The effect of the intervention on the severity of Anxiety and Depression. The total score for each subscale of the HADS ranges from 0 to 21 with higher score indicates more severe anxiety or depression (worse).
The Quality of Life (using Medical Outcomes Study Short Form 12) | 2 months post intervention.
  The effect of the intervention on Quality of Life. The total score ranges between 0% to 100% with higher score indicates a better quality of life (better).
Cognitive ability (using Montreal Cognitive Assessment) | 2 months post intervention.
  The effect of the intervention on Cognitive ability. The total score ranges from 0 to 30 points with a score of 25 or less indicating cognitive impairment (worse).

CONTACTS AND LOCATIONS:
Overall Officials: Alia A Alghwiri, Principal Investigator — University of Jordan
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT04818008/SAP_000.pdf